CLINICAL TRIAL: NCT01090947
Title: Data Aquisition for Optimization of Coronary Artery Disease Algorithm
Status: Completed | Type: Observational
Sponsor: Acarix (Industry)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: CP002IN
Record Dates: First submitted 2010-03-18; First posted 2010-03-23 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients referred to CAG.: Sequential design with ProtoCAD and CAG
  Interventions: Device: ProtoCAD

INTERVENTIONS:
Device: ProtoCAD — Aquiring acoustic signals from heart patients.
  Other Names: Acarix CAD device.

SUMMARY:
The purpose of the study is to optimize an already existing algorithm for diagnosing atherosclerosis of the coronary arteries (CAD, Coronary Artery Disease).

DETAILED DESCRIPTION:
Acoustic information from the heart is obtained from patients suffering from Coronary Artery Disease. The acoustic signals are evaluated as indicators for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum 18 years
* Referred to CAG on suspicion of CAD
* Stabile angina without ACS
* Signed informed consent

Exclusion Criteria:

* ACS
* Previous bypass operation
* Previous heart transplant(incl. mechanical or artificial)
* Pregnancy
* Damaged skin on examination location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to CAG.
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Sensitivity versus 1-specificity as a function of cut-off values on the 'Cardiac Noise Marker' scale here under Sensitivity by suitable cut-off value on the 'Cardiac Noise Marker' scale and Specificity with same cut-off value. | The first testday

SECONDARY OUTCOMES:
Observed differences in distribution of 'Cardiac Noise Marker' within three sub-groups. | The first testday

CONTACTS AND LOCATIONS:
Overall Officials: Peter Clemmensen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University Hospital of Copenhagen, Copenhagen, Denmark